CLINICAL TRIAL: NCT02215486
Title: Head Massage Intervention to Decrease Physiological Signs of Stress as Assessed by Changes in the Autonomic Nervous System Functions in Healthy Volunteers: A Pilot Study
Brief Title: The Effect of Head Massage Therapy on the Regulation of the Autonomic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's & Women's Health Centre of British Columbia (Other)
Responsible Party: Principal Investigator, Jean-Paul Collet, Director, Children's & Women's Health Centre of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H13-03391
Record Dates: First submitted 2014-08-09; First posted 2014-08-13 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: The Effect of Head Massage Therapy on the Autonomic Nervous System
Keywords: Head massage therapy; Massage therapy; Autonomic nervous system (ANS); Heart rate variability (HRV); Pre-ejection period (PEP)

INTERVENTIONS:
Other: Head Massage Therapy — Intervention consists of administering head massage therapy according to the Chinese head massage protocol for approximately 10 minutes.
Other: Simple relaxation (No Head Massage) — Consists of a simple relaxation in the same sitting position as the head massage therapy session.

SUMMARY:
The autonomic nervous system (ANS) unconsciously regulates the activities of vital organ systems such as the respiratory, circulatory, and urinary systems. It consists of two major components, the parasympathetic nervous system (PNS) and the sympathetic nervous system (SNS), which together are in charge of keeping our body in homeostasis. Homeostasis is the state of chemical and metabolic balance within an organism; it is disturbed in situations of uncontrolled stress.

Massage has been shown to decrease SNS and stimulate PNS; but most studies focused on full body massage, with limited assessment of ANS function, and lacked control groups.

The effects of head massage therapy (HMT) on regulating the activity of the ANS have not been studied before. In this pilot study, we propose that by randomizing 10 participants to sessions of HMT and 'Simple Relaxation' (no HMT), and by using a non-invasive method of measuring the ANS activity (spectral analysis of Heart Rate Variability [HRV] as well as Pre-ejection Period (PEP)), we will be able to investigate the effects of 10 minutes of HMT in comparison with the period of no HMT administered. We expect HMT to reduce stress, with a better and balanced profile of autonomic nervous system after receiving massage.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy individuals

Exclusion Criteria:

* Use of anti-depressants or drugs that affect the cardiovascular system or ANS
* Smoking more than 10 cigarettes/day
* Inability to provide consent
* Inability to speak and/or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) parameters | Within 1 day
  Main HRV parameters that will be reported include High Frequency (HF) which is the power in high frequency range representative of the parasympathetic nervous system activity, HFnu which is the HF power in normalized units, and total power which is the total variability of the autonomic nervous system over the temporal segment.
  HRV parameters are measured at baseline and post intervention. Post-intervention outcomes for each subject will be compared with their baseline. There will also be comparison of the outcomes between the massage and the control intervention, for the effect of massage therapy
Pre-ejection period (PEP) | Within 1 day
  PEP is the time interval between electrical stimulation of the sinoatrial node and opening of the aortic valves and has shown to be inversely correlated with the activity of the sympathetic nervous system.
  PEP is measured at baseline and post intervention. Post-intervention outcomes for each subject will be compared with their baseline. There will also be comparison of the outcomes between the massage and the control intervention, for the effect of massage therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Collet, MD, PhD, Principal Investigator — Children's & Women's Health Centre of British Columbia; Mir Sohail Fazeli, M.D., Principal Investigator — The University of British Columbia
Locations (1):
- BC Children's and Women's Hospital, Vancouver, British Columbia, Canada